CLINICAL TRIAL: NCT05559294
Title: Effect of Professional Development in Science for Early Childhood Education and Care Staff
Brief Title: Effect of Professional Development in Science
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: UCL University College, Denmark (Other)
Collaborators: VIVE - The Danish Center for Social Science Research (Other)
Responsible Party: Principal Investigator, Tine Nielsen, Associate Professor, UCL University College, Denmark
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: STB Trial 9012102
Record Dates: First submitted 2022-09-21; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Early childhood education and care; Early childhood educators; Self-efficacy for science; Attitudes toward science; Engagement with science; Professional development; Science capital
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional development (Experimental): The intervention consists of a nine months long professional development program with an interchange between three e-learning modules and three group workshops starting with an e-learning module and ending with a workshop. Each workshop is 3 hours with approximately 100 participants. The e-learning modules are completed individually by ECEC staff. Between workshops, each day nursery and/or kindergarten center will receive a two-hour supervisory visit from UCL staff to support professional development. The daily leader at the day nursery and/or kindergarten center sets the theme for each supervisory visit to enhance development as much as possible.
  The intervention is being designed as a collaboration between UCL and Odense municipality
  Interventions: Behavioral: Professional Development of Early Childhood Education and Care Staff for Science
- Usual professional development (Active Comparator): Education and Care as Usual entails a standing offer from the municipality of Odense for Usual Competence development within the area of nature, outdoor life and natural phenomena visits from a learning consultant to support the ECEC staff's work with digital technology at the day nursery and/or kindergarten center. It is up to the day nursery and/or kindergarten center if the use the offer or not. This offer is extended to all day nursery and/or kindergarten centers.
  Interventions: Behavioral: Education and care as Usual (ECAU)

INTERVENTIONS:
Behavioral: Professional Development of Early Childhood Education and Care Staff for Science — A nine-month program consisting of three e-learning modules and three group workshops
  Arms: Professional development
Behavioral: Education and care as Usual (ECAU) — Active control
  Arms: Usual professional development

SUMMARY:
This trial is a randomized controlled trial aimed at assessing the effectiveness of a nine-month-long professional development program to improve early childhood educators' and carers' self-efficacy for science approaches, engagement with science, and attitudes toward science in early childhood education and care (ECEC).

DETAILED DESCRIPTION:
Early childhood education and care (ECEC) staff often struggle in working with science with small children, as the National Strengthened Pedagogical Curriculum (Ministry of Children and Education, 2020) is difficult to put into practice. Thus, they are challenged with regard to meeting the national objectives for this in this regard. A large-scale professional development program is developed and implemented to overcome this gap and to enhance ECEC staff's self-efficacy, engagement with, and attitudes toward science.

The intervention is developed by UCL teaching staff in collaboration with the municipality of Odense with the aim of offering all children in Odense municipality's ECEC program a playful and investigative approach to science as defined in the national curriculum theme 'Nature, outdoor life and natural phenomena' by offering ECEC staff extensive professional development in this field. The professional development course will be delivered by UCL teaching staff from the area of early childhood education and care in two consecutive runs, each of nine months duration.

The professional development consists of a combination of three workshops and three e-learning modules. In between workshops and e-learning modules, the ECEC staff implement the content practically by working with science with the children, while receiving supervision from a teacher from the professional development. The set-up is based on the model of teacher professional growth (Clark & Hollingsworth, 2002). The aim of the professional development program is that ECEC staff becomes able to construct and enhance science-oriented learning environments, thus providing the children with educative experiences with science (Dewey, 1913). The aim of the trial is to assess the effectiveness of the intervention to improve early childhood educators' and carers' self-efficacy for science approaches, engagement with science, and attitudes toward science in early childhood education.

The study is a Randomized Controlled Trial (RCT). A total of approximately 1400 ECEC staff will be randomized to the professional development in the first run or Education and Care as Usual (ECAU). The ECAU group in the first run will receive the intervention in a second run once the first run is completed.

Participants are ECEC staff in pedagogical positions (i.e. pedagogues, assistants, assistant teachers, and daily leaders) employed in a combined nursery and kindergarten in Odense municipality. Participants must be able to fill out questionnaires in Danish.

Data will be collected at baseline (pre-intervention), after 4.5 months (midway), and 9 months after baseline, when the intervention is completed.

ELIGIBILITY:
Inclusion Criteria:

* Adults employed in a day nursery and/or kindergarten center in the municipality of Odense at the start of the intervention
* Employed in one of four pedagogical positions: pedagogues [pædagoger], assistants [pædagogiske assistenter], assistant teachers [pædagogmedhjælpere], and daily leaders [dalig leder]

Exclusion Criteria:

* Employed in other positions than the four above in a day nursery and/or kindergarten center
* "at home child carers" [dagpleje]
* Not able to fill out questionnaires in Danish

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change in Self-efficacy for science approach at 4.5 months | Baseline, 4,5 months
  Self-Efficacy for Science Approach (SESA) in early childhood educators and carers. The scale will be developed for purpose with a basis in the National Strengthened Pedagogical Curriculum prior to baseline. Rasch measurement models will be used for validation, including analyses of differential item functioning to ensure that the two groups of staff in the RCT can be compared unbiased. The resulting scale will consist of approximately 15 items (score range 0-60) and have sufficient reliability.
  Higher scores are better.
Change in Self-efficacy for science approach at 9 months | Baseline, 9 months
  Self-Efficacy for Science Approach (SESA) in early childhood educators and carers. The scale will be developed for purpose with a basis in the National Strengthened Pedagogical Curriculum prior to baseline. Rasch measurement models will be used for validation, including analyses of differential item functioning to ensure that the two groups of staff in the RCT can be compared unbiased. The resulting scale will consist of approximately 15 items (score range 0-60) and have sufficient reliability.
  Higher scores are better.

SECONDARY OUTCOMES:
Science capital for professionals | Baseline
  The inventory was adapted from the STEM Capital questionnaire developed from the ESRC-funded ASPIRES study at University College London (https://www.ucl.ac.uk/ioe/departments-and-centres/departments/education-practice-and-society/aspires-research) designed for adult higher education students to achieve questions aimed at early childhood educators and carers. For the Attitudes towards Science subscale, some items were also adapted from the Science attitude scales developed by Francis & Greer (1999) and Oon et al (2019).
  The SCPI consist of three subscales and three single item questions, which form the Science Capital for Professionals construct.
  * Attitudes towards Science Scale (ASS)
  * Engagement with Science in the Work context (ES-work)
  * Engagement with in the non-work context (ES-life)
  * Three single items on aspects of relationship with science The total SCPI instrument consist of 57 items, range 0-100 (lowest value in each item scored as zero), higher is better.
Change in Attitudes toward science at 4.5 months | Baseline, 4,5 months
  Attitudes towards Science Scale (ASS) from the Science Capital for Professional Inventory (SCPI), 10 items, range 0-20, higher is better.
Change in Attitudes toward science at 9 months | Baseline, 9 months
  Attitudes towards Science Scale (ASS) from the Science Capital for Professional Inventory (SCPI), 10 items, range 0-20, higher is better.
Change in engagement with science in the work life at 4.5 months | Baseline, 4,5 months, 9 months
  Engagement with Science in the Work context subscale (ES-work) from the Science Capital for Professional Inventory (SCPI), 17 items, range 0-36, higher is better.
Change in engagement with science in the work life at 9 months | Baseline, 9 months
  Engagement with Science in the Work context subscale (ES-work) from the Science Capital for Professional Inventory (SCPI), 17 items, range 0-36, higher is better.
Motivation for professional development in science | Baseline
  Expectancy-value Motivation for Engaging in Professional Development in Science (EMEPDS). The inventory will be adapted to the target group from the Expectancy-Value-Cost Scale for students (Kosovich et al., 2015), 10 items, range 0-30. Higher is better
science approach behaviors | 9 months
  Practicing Science Scale (PSS). The scale assesses context-specific ECEC staff behaviors indicating a pedagogical approach implementing the National Strengthened Pedagogical Curriculum objectives with regard to science and technology, 5 items, range 0-15. Higher is better.

CONTACTS AND LOCATIONS:
Overall Officials: Morten R petersen, PhD, Study Director — UCL University college
Locations (1):
- UCL university college, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared on request and will consist of the primary outcome data as well as secondary measures and background information, as necessary to re-analyse.
Time Frame: Data will become available once we have published study protocol, validation study on the primary outcome, and study report. Expected that this will be possible by the start of 2026 and two years forward.
Access Criteria: purpose of data request as re-analyses using alternative methods.

REFERENCES:
- [Background] Clarke D, Hollingsworth H. Elaborating a model of teacher professional growth. Teaching and teacher education. 2002; 18(8): 947-967.
- [Background] Dewey J. Interest and effort in education.1913. Boston, MA, US: Houghton, Mifflin and Company.
- [Background] Francis LJ, Greer JE. Measuring Attitude Towards Science Among Secondary School Students: the affective domain. Research in Science & Technological Education. 1999; 17(2): 219-226.
- [Background] Kosovich JJ, Hulleman CS, Barron KE, Getty S. A Practical Measure of Student Motivation: Establishing Validity Evidence for the Expectancy-Value-Cost Scale in Middle School. The Journal of Early Adolescence. 2015; 35(5-6):790-816.
- [Background] Oon P-T, Hu BY, We B. Early childhood educators' attitudes toward science teaching in Chinese schools. Australasian Journal of Early Childhood. 2019; 44(4): 423-435.
- See also: the ESRC-funded ASPIRES study at University College London — https://www.ucl.ac.uk/ioe/departments-and-centres/departments/education-practice-and-society/aspires-research